CLINICAL TRIAL: NCT00507403
Title: Effect of Methotrexate on the Relation Dose-effect of Infliximab in Ankylosing Spondylitis
Brief Title: Infliximab and Methotrexate in Ankylosing Spondylitis
Acronym: SPAXIM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PHRR/04/PG-SPAXIM
Record Dates: First submitted 2007-07-24; First posted 2007-07-26 (Estimated); Last update posted 2017-01-16 (Estimated); Status verified 2017-01

CONDITIONS: Ankylosing Spondylitis
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Infliximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Infliximab (Active Comparator): Infliximab
  Interventions: Drug: infliximab
- Infliximab +methotrexate (Experimental): Infliximab +methotrexate
  Interventions: Drug: infliximab

INTERVENTIONS:
Drug: infliximab

SUMMARY:
There is a great individual variability of pharmacokinetic of infliximab in patients treated for ankylosing spondylitis (AS). Moreover, some patients have a treatment with methotrexate (MTX), others have not.

Thus, the aim of this study is to assess the effect of MTX on the pharmacokinetic properties of infliximab in 30 patients treated for AS, 15 with MTX, 15 without.

ELIGIBILITY:
Inclusion Criteria:

* Ankylosing spondylitis
* Needing anti-TNF drugs

Exclusion Criteria:

* Contra-indications to anti-TNF drugs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-10; Primary Completion 2009-10 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic properties of infliximab in AS patients with or without methotrexate | 16 weeks

SECONDARY OUTCOMES:
Individual pharmacokinetic modelisation of infliximab | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: PHILIPPE GOUPILLE, MD, Principal Investigator — University hospital of Tours, France
Locations (2):
- France (2):
  - University Hospital Jean MINJOZ -Besançon, Besançon
  - University hospital of Tours, Tours

REFERENCES:
- [Derived] Mulleman D, Lauferon F, Wendling D, Ternant D, Ducourau E, Paintaud G, Goupille P. Infliximab in ankylosing spondylitis: alone or in combination with methotrexate? A pharmacokinetic comparative study. Arthritis Res Ther. 2011 Jun 3;13(3):R82. doi: 10.1186/ar3350. PMID 21639907